CLINICAL TRIAL: NCT06009887
Title: The Effect of Motivational Interviews of Primiparous Pregnants With Low Belief in Normal Birth on Medical and Natural Birth Beliefs
Brief Title: Motivational Interview in Primiparous Pregnants With Low Belief in Normal Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Çiğdem KARAKAYALI AY, PhD Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/1198
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Natural birth belief; Medical birth belief; Motivational interview.
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: İntervention Group (Experimental): Motivational interviewing is a counseling approach that pays special attention to the language of change, adopts a collaborative, goal-oriented communication style and aims to strengthen personal motivation and commitment to this change, revealing and discovering the reasons for the change in one's own, in an atmosphere of acceptance and empathy.
  Interventions: Behavioral: Motivational Interview
- No Intervention: Control Group (No Intervention): No interventions were made for those in the control group other than routine hospital practices.

INTERVENTIONS:
Behavioral: Motivational Interview — Motivational interviewing is a collaborative speaking style to strengthen one's own motivation and commitment to change. Motivational interviewing is not a technique but a fundamental therapeutic style that does not try to make people change their behavior against their will. Proven to be effective in many areas of healthcare, motivational interviewing is widely used to help people resolve their indecision about change, explore their concerns, and set their own goals. The purpose of the motivational interviews conducted in the study is to increase the belief in normal and natural birth by enabling pregnant women to understand the factors that affect their low belief in normal birth, to take action for change and to believe in change, and to minimize the practices that cause medicalization of birth such as cesarean section by reducing medical birth beliefs.
  Arms: Experimental: İntervention Group

SUMMARY:
This study aims to determine the effect of motivational interviews made with primiparous pregnant women with low belief in normal birth on medical and natural birth belief. This randomized controlled study was conducted in a randomized controlled manner with a total of 148 pregnant women who applied to the obstetrics outpatient clinic of a hospital in eastern Turkey (74 trials, 74 controls). In the study, a total of four sessions of motivational interviews were conducted with the primiparous pregnant women in the experimental group, one week apart. No intervention was applied to the women in the control group. Research data Personal Information Form, Belief Scale for Normal Delivery (BSND) and Birth Beliefs (Natural and medical birth belief) Scale (BBS) were used. Descriptive statistics, Pearson's chi-square test, and dependent and independent t-test were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Having a low level of belief and tendency towards normal birth according to the Normal Birth Belief Scale (between 24-56 points),
* Primiparous pregnant,
* According to the calculations made by USG of the pregnant women who do not know the last menstruation date or the last menstruation date, 24-36 days of pregnancy. in the week,
* Pregnant women who volunteered were included in the sample of the study.

Exclusion Criteria:

* Premature birth,
* Having any risk diagnosed during pregnancy (such as preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios),
* Contraindications for normal vaginal delivery
* Developing cesarean indication,
* Not completing MG sessions,
* Pregnant women with deficiencies or errors in any of the forms in which the data were obtained were excluded from the sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Belief Scale for Normal Delivery (BSND) | up to 4 weeks
  It was developed to evaluate the beliefs and tendencies of pregnant women towards normal birth. The scale is a five-point Likert type and is scored as I completely agree (5), agree (4), undecided (3), disagree (2), strongly disagree (1). A minimum of 24 and a maximum of 120 points can be obtained from the scale. If the total score from the scale is between 24 and 56, low, between 57 and 88, moderate, and between 89 and 120, high-level beliefs and tendency towards normal birth are in question. As the average score obtained from the scale increases, the beliefs and tendencies of pregnant women about normal birth increase.
Birth Beliefs (Natural and medical birth belief) Scale (BBS) | Baseline and 4 weeks
  While one of the sub-dimensions of the scale used to evaluate the basic belief levels of women about childbirth evaluates birth as a natural process, the other sub-dimension considers birth as a medical/medical process. The scale consists of 11 items in total, including 5 items (items 3, 5, 7, 8, and 11) for the belief in the natural process of birth and 6 items (items 1, 2, 4, 6, 9, and 10) for the belief in the medical/medical process. consists of. The scale score is obtained by dividing the total score of the items belonging to each sub-dimension by the number of items belonging to that sub-dimension. The group with a high numerical value in the arithmetic mean result constitutes the birth belief of the woman. In this Likert-type scale, each item is scored between 1 and 5 scales. The option "strongly disagree" receives 1 point, while the option "strongly agree" receives 5 points.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem KARAKAYALI AY, Principal Investigator — Department of Midwifery, Faculty of Health Sciences, Sutcuimam University
Locations (1):
- Department of Midwifery, Faculty of Health Sciences Sutcuimam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. Because the institution where the research was conducted does not allow this.

REFERENCES:
- [Result] Rasouli M, AtashSokhan G, Keramat A, Khosravi A, Fooladi E, Mousavi SA. The impact of motivational interviewing on participation in childbirth preparation classes and having a natural delivery: a randomised trial. BJOG. 2017 Mar;124(4):631-639. doi: 10.1111/1471-0528.14397. Epub 2016 Nov 10. PMID 27862837
- See also: The impact of motivational interviewing on participation in childbirth preparation classes and having a natural delivery: a randomised trial — https://pubmed.ncbi.nlm.nih.gov/27862837/